CLINICAL TRIAL: NCT00088491
Title: A Double-Blind, Randomized Study Comparing Intramuscular Olanzapine Depot to Oral Olanzapine and Low-Dose Depot in the Maintenance Therapy of Patients With Schizophrenia
Brief Title: Comparison of Intramuscular Olanzapine Depot to Oral Olanzapine and Low-Dose Depot in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5985; F1D-MC-HGKA
Record Dates: First submitted 2004-07-26; First posted 2004-07-28 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Schizophrenic Disorders
MeSH Terms: conditions — Schizophrenia | interventions — Olanzapine

INTERVENTIONS:
Drug: Intramuscular Olanzapine Depot
Drug: Oral Olanzapine

SUMMARY:
This is a randomized, double-blind study to determine how well intramuscular (IM) olanzapine depot works compared to oral olanzapine; evaluate the safety and tolerability of IM olanzapine depot compared to oral olanzapine; evaluate different doses of IM olanzapine depot; and determine the blood levels of IM olanzapine depot in patients at different points in time after an injection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have schizophrenia
* Patients must be clinically stable on antipsychotic medication
* Patients must be retrospectively judged by investigators, based on clinical interview and impression, to have been stable (with respect to their symptoms of schizophrenia) for at least 4 weeks entry into the study
* Patients must be an outpatient and have BPRS positive items scores of 4 or less to enter the study
* Female patients of childbearing potential must be using a medically accepted means of contraception.

Exclusion Criteria:

* Patients must not have participated in a clinical trial of another investigational drug, including olanzapine, within 1 month (30 days) prior to study entry.
* Female patients must not be pregnant or breast-feeding
* Patients must not be experiencing acute, serious, or unstable medical conditions other than schizophrenia
* Patients must not require concomitant treatment with any other medication with primarily central nervous system activity, including antidepressants, mood stabilizers, and anticonvulsants.
* Patients must not have a substance (except nicotine or caffeine) dependence within the past 30 days

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1205 (Actual)
Dates: Start 2004-06; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Determine comparative efficacy in patients with schizophrenia of non-inferiority of IM olanzapine depot high and low doses versus oral olanzapine based on exacerbation rates after 6 months of maintenance treatment
Determine comparative efficacy in patients with schizophrenia of superiority of IM olanzapine depot low, med and high doses versus very low dose based on time to exacerbation of symptoms of schizophrenia

SECONDARY OUTCOMES:
Demonstrate non-inferior efficacy in terms of exacerbation rates of high plus low dose IM olanzapine depot versus medium dose
Provide information on transition of patients stabilized on oral olanzapine 10, 15 or 20 mg/day to therapeutic doses of IM olanzapine depot
Demonstrate superiority of high dose, medium dose and low dose IM olanzapine depot compared with very low dose IM olanzapine depot in change from baseline to endpoint in PANSS total, positive, negative and general subscales
Assess the safety and tolerability of high plus low dose IM olanzapine depot versus oral olanzapine
Assess the safety and tolerability of medium dose IM olanzapine depot versus oral olanzapine
Assess the safety and tolerability of each IM olanzapine depot treatment group versus very low dose IM olanzapine depot
Compare the efficacy of high plus low dose IM olanzapine depot versus oral olanzapine during maintenance treatment on quality of life, drug attitude inventory, resource utilization and hospitalization measures
Compare the efficacy of high, medium and low doses of IM olanzapine depot during maintenance treatment on quality of life, drug attitude inventory, resource utilization and hospitalization measures
Characterize the pharmacokinetics of olanzapine following multiple dosing with IM olanzapine depot at each of the prescribed dosing regimens and to compare IM olanzapine depot pharmacokinetics with oral olanzapine pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pitkäniemi, Finland
- Turkey (Türkiye) (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ankara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Istanbul
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Izmir

REFERENCES:
- [Derived] Atkins S, Detke HC, McDonnell DP, Case MG, Wang S. A pooled analysis of injection site-related adverse events in patients with schizophrenia treated with olanzapine long-acting injection. BMC Psychiatry. 2014 Jan 14;14:7. doi: 10.1186/1471-244X-14-7. PMID 24423017
- [Derived] Ascher-Svanum H, Novick D, Haro JM, Bertsch J, McDonnell D, Detke H. Predictors of psychiatric hospitalization during 6 months of maintenance treatment with olanzapine long-acting injection: post hoc analysis of a randomized, double-blind study. BMC Psychiatry. 2013 Sep 16;13:224. doi: 10.1186/1471-244X-13-224. PMID 24041270
- [Derived] Peuskens J, Porsdal V, Pecenak J, Handest P, D'yachkova Y, Brousil R, Deberdt W. Schizophrenia symptoms and functioning in patients receiving long-term treatment with olanzapine long-acting injection formulation: a pooled analysis. BMC Psychiatry. 2012 Aug 31;12:130. doi: 10.1186/1471-244X-12-130. PMID 22935168
- [Derived] McDonnell DP, Kryzhanovskaya LA, Zhao F, Detke HC, Feldman PD. Comparison of metabolic changes in patients with schizophrenia during randomized treatment with intramuscular olanzapine long-acting injection versus oral olanzapine. Hum Psychopharmacol. 2011 Aug;26(6):422-33. doi: 10.1002/hup.1225. Epub 2011 Aug 5. PMID 21823172
- [Derived] Hill AL, Sun B, Karagianis JL, Watson SB, McDonnell DP. Dose-associated changes in safety and efficacy parameters observed in a 24-week maintenance trial of olanzapine long-acting injection in patients with schizophrenia. BMC Psychiatry. 2011 Feb 15;11:28. doi: 10.1186/1471-244X-11-28. PMID 21324135
- [Derived] McDonnell DP, Detke HC, Bergstrom RF, Kothare P, Johnson J, Stickelmeyer M, Sanchez-Felix MV, Sorsaburu S, Mitchell MI. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, II: investigations of mechanism. BMC Psychiatry. 2010 Jun 10;10:45. doi: 10.1186/1471-244X-10-45. PMID 20537130
- [Derived] Detke HC, McDonnell DP, Brunner E, Zhao F, Sorsaburu S, Stefaniak VJ, Corya SA. Post-injection delirium/sedation syndrome in patients with schizophrenia treated with olanzapine long-acting injection, I: analysis of cases. BMC Psychiatry. 2010 Jun 10;10:43. doi: 10.1186/1471-244X-10-43. PMID 20537128
- [Derived] Kane JM, Detke HC, Naber D, Sethuraman G, Lin DY, Bergstrom RF, McDonnell D. Olanzapine long-acting injection: a 24-week, randomized, double-blind trial of maintenance treatment in patients with schizophrenia. Am J Psychiatry. 2010 Feb;167(2):181-9. doi: 10.1176/appi.ajp.2009.07081221. Epub 2009 Dec 15. PMID 20008947
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com